CLINICAL TRIAL: NCT01044823
Title: Use of Thermal and 3D Imaging to Quantify Arthritis
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO08040135; R21AR056690 (NIH)
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2011-02

CONDITIONS: Rheumatoid Arthritis; Juvenile Rheumatoid Arthritis
Keywords: RA; JRA
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult RA
  Interventions: Other: 3D and thermal imaging
- pediatric JRA
  Interventions: Other: 3D and thermal imaging

INTERVENTIONS:
Other: 3D and thermal imaging — subjects will be imaged before and after receiving DMARD therapy

SUMMARY:
One of the biggest challenges in caring for patients with Rheumatoid Arthritis (RA) and Juvenile Rheumatoid Arthritis (JRA) is quantifying the degree of disease activity in any given joint. We have built a prototype device using well-established sensors to rapidly quantify surface swelling and heat in arthritic joints. The goal of our studies is to test the hypothesis that this Imager can improve the clinical assessment of arthritis.

ELIGIBILITY:
Inclusion Criteria:

* at least 4 years of age

Exclusion Criteria:

* less than 4 years of age

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with JRA adults with RA
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States